CLINICAL TRIAL: NCT03301116
Title: Promoting Seniors' Health With Home Care Aides: A Randomized Controlled Trial
Brief Title: Promoting Seniors' Health With Home Care Aides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Naoko Muramatsu, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0689; R01AG053675 (NIH)
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Muscle Weakness
Keywords: Exercise; Frail Elderly; Homebound Persons; Activities of Daily Living; Mobility Limitation; Home Care Services; Long-Term Care; Dual MEDICAID MEDICARE Eligibility
MeSH Terms: conditions — Muscle Weakness; Motor Activity; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Home care aide-client pairs will be randomly assigned to one of two groups in parallel for the duration of the study. Home care aides will not be allowed to have multiple participating clients assigned to different groups to prevent group contamination.
Who Masked: Outcomes Assessor
Masking Description: N/A (there are no other parties who will be masked in the clinical trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Moves (Experimental): Home care aides (HCAs) will be trained to deliver Healthy Moves for Aging Well (Healthy Moves), a gentle physical activity program, to their clients. On the first home care visit after the training, HCAs will introduce the program, assess their clients' readiness for the activity and have their clients set personally meaningful goals, and teach the three chair-bound moves. Home care clients will be asked to do the three moves every day. HCAs remind clients of their activity as part of their regular home care visits throughout the 4-month intervention period.
  Interventions: Behavioral: Healthy Moves for Aging Well (Healthy Moves)
- Active Mind (Active Comparator): Home care aides (HCAs) will be trained to deliver Active Mind for Aging Well (Active Mind), a gentle thinking activity program, to their clients. On the first home care visit after the training, HCAs will introduce the program, assess their clients' readiness for the activity and have their clients set personally meaningful goals, and teach the activity. Home care clients will be asked to do a word search puzzle every day. HCAs remind clients of their activity as part of their regular home care visits throughout the 4-month intervention period.
  Interventions: Behavioral: Active Mind for Aging Well (Active Mind)

INTERVENTIONS:
Behavioral: Healthy Moves for Aging Well (Healthy Moves) — A safe physical activity program which consists of a brief motivational enhancement and three movements to be performed in a seated position. The intervention will be delivered by home care aides for their clients.
  Arms: Healthy Moves
Behavioral: Active Mind for Aging Well (Active Mind) — A word puzzle program which consists of a brief motivational enhancement and word search activities. The intervention will be delivered by home care aides for their clients.
  Arms: Active Mind

SUMMARY:
This study aims to test whether a safe physical activity program with a built-in motivational enhancement component, performed in a seated position, preserves the function and well-being of older home care clients.

DETAILED DESCRIPTION:
Regular physical activity benefits older adults physically and mentally. However, the availability and the evidence for physical activity programs that are safe and appropriate for home-bound older adults at risk for nursing home admission are limited. The current project aims to examine the effectiveness of a safe physical activity program, led by home care aides who regularly help hard-to-reach older home care clients with housekeeping and routine personal care services in the home. The primary aim is to test whether the safe physical activity program with a built-in motivational enhancement component, performed in a seated position, preserves the function and well-being of home care clients. The secondary aim is to understand for whom the program is efficacious, the extent to which the program can reach the target population, the extent to which participants drop out of the program, the extent to which program participants maintain the behavioral change introduced by the intervention, and what the program's cost-effectiveness is. Building on a pilot project that demonstrated the program's feasibility in a large home care program funded by the state and Medicaid, this randomized controlled trial will inform future expansion of the physical activity program into real-world home care settings.

ELIGIBILITY:
HOME CARE CLIENTS

Inclusion Criteria:

* English or Spanish-speaking older adults aged 60+
* Receiving Illinois Department on Aging Community Care Program In-Home service from the collaborating home care agency
* Able to sit in a chair independently for >=15 minutes (it is fine if the person needs help with transferring to a chair)
* Cognitive status sufficient to follow directions and respond to survey questions as determined by the Six-Item Screener (Callahan, et al., 2002) (the instrument used in the phone screening) and the Modified Mini-Mental State (3MS) Examination (the instrument used in the in-home screening)
* Willing to be assigned to either intervention program
* Willing to have the research team notify the primary care physician of the client's study participation

Exclusion Criteria:

* Having a legal guardian appointed
* Bedridden or unable to sit in a chair independently
* Receiving hospice care or having a terminal diagnosis
* Self-reported inability to read large print books

HOME CARE AIDES

Inclusion Criteria:

* English or Spanish-speaking home care aide caring for an older home care client eligible for the study
* Age 18 and older
* Willing to implement the intervention program routine with their eligible client(s) for the full 4 months
* Willing to be randomly assigned to either intervention program
* Intend to be a home care aide for the next 12 months

Exclusion Criteria

• Not having a home care client who participates in the study

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Function (Daily activity difficulties and dependency in older home care clients) at Month 4 | Month 4
  Activities of daily living that are specifically targeted by the intervention (6-items scale; each task will be scored 0-no difficulty/no help; 1=difficulty but no help; 2=need help; summed score, range 0-12)

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline, Month 4, Month 8
  Range 0-12 (Guralnik et al., 1994)
Exercise-related social support from home care aides | Baseline, Month 4, Month 8
  Frequency of support from home care aides. Three items, range 3-9. Adapted from Sallis et al. (1987)
Self-rated health | Baseline, Month 4, Month 8
  General self-rated health, range 1-5 (poor to excellent)
Fear of falling | Baseline, Month 4, Month 8
  Short Falls Efficacy Scale-International (FES-I), seven items, 4-point scale (not at all worried to very worried), range 7-28 (Kempen et al., 2008).

OTHER OUTCOMES:
Basic activities of daily living (secondary outcome) | Baseline, Month 4, Month 8
  8-item scale; each task will be scored 0-no difficulty/no help; 1=difficulty but no help; 2=need help, summed score range 0-16 (Gill, Robinson, and Tinetti, 1998)
Activities of daily living that are specifically targeted by the intervention (secondary outcome) | Baseline, Month 4, Month 8
  6-item scale; each task will be scored 0-no difficulty/no help; 1=difficulty but no help; 2=need help, summed score range 0-12
Instrumental activities of daily living (secondary outcome) | Baseline, Month 4, Month 8
  4-item scale; each task will be scored 0-no difficulty/no help; 1=difficulty but no help; 2=need help, summed score range 0-8
Physical activity levels (secondary outcome) | Baseline, Month 4, Month 8
  Days and amount of time spent on three types of physical activity in the past week: strengthening, stretching, and aerobics
Falls (secondary outcome) | Baseline, Month 4, Month 8
  Number of falls in the past 4 months, and whether any reported falls led to injury that needed medical attention (Yes/No)
Ankle range of motion (secondary outcome) | Baseline, Month 4, Month 8
  Angle between ankle dorsiflexion and plantarflexion in degrees
Pain (secondary outcome) | Baseline, Month 4, Month 8
  A scale adapted from SF36 to measure pain, after taking pain medication if applicable, range 0-10
Depressive symptoms (secondary outcome) | Baseline, Month 4, Month 8
  Feelings in the past week. 9-item scale (Yes/No), range 0-9

CONTACTS AND LOCATIONS:
Overall Officials: Naoko Muramatsu, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
After the end of the study, data collection instruments, codebooks, and other data documentation will be made available in conjunction with the dataset in a standard format that is readable across a variety of applications. Guidelines from relevant state agencies and collaborators will be followed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the main study results
Access Criteria: To protect participants from re-identification while retaining the analytic utility of the data, the data and associated documentation will be available to users only under a data-sharing agreement, managed by the National Archive of Computerized Data on Aging (NACDA), that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will only be released once all Institutional Review Board (IRB) approvals and human subjects concerns have been addressed.